CLINICAL TRIAL: NCT02221999
Title: A Prospective, Randomized, Open-label Comparison of Preoperative Weekly Paclitaxel and Cisplatin With or Without Endocrine Therapy in Patients With Operable Hormone Receptor Positive and Triple Negative Locally Advanced Breast Cancer
Brief Title: Weekly Paclitaxel and Cisplatin to Treat Hormone Receptor Positive and Triple Negative Breast Cancer Patients
Acronym: SHPD002
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Lu, professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-BC-002
Record Dates: First submitted 2014-07-14; First posted 2014-08-21 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Tubular Breast Cancer; Mucinous Breast Cancer; Invasive Ductal Breast Cancer; Inflammatory Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — Paclitaxel; Cisplatin; Gonadotropin-Releasing Hormone; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chemotherapy only (Active Comparator): Paclitaxel injection 80mg/m2,given on days1,8,15 and 22 of a 28-day cycle；Cisplatin 25mg/m2, given on days 1,8,and 15 of a 28-day cycle； for 4 cycles
  Interventions: Drug: Paclitaxel; Drug: Cisplatin
- GnRHa (Experimental): Paclitaxel 80mg/m2,given on days1,8,15 and 22 of a 28-day cycle; Cisplatin 25mg/m2, given on days 1,8,and 15 of a 28-day cycle; for 4 cycles Gonadotropin-releasing hormone agonist （GnRHa）11.25 mg every 3 months or 3.6mg every month subcutaneously
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Gonadotropin-releasing hormone agonist
- letrozole (Experimental): Paclitaxel 80mg/m2,given on days1,8,15 and 22 of a 28-day cycle; Cisplatin 25mg/m2, given on days 1,8,and 15 of a 28-day cycle; for 4 cycles Letrozole 2.5mg/day
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Letrozole

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
Drug: Cisplatin
Drug: Gonadotropin-releasing hormone agonist — Goserelin 3.6 mg q28d or Leuprolide 11.25 mg q3m
  Arms: GnRHa
Drug: Letrozole
  Arms: letrozole

SUMMARY:
The investigators hypothesize that paclitaxel combined with cisplatin in a weekly-based regimen as neoadjuvant chemotherapy is effective and tolerable for locally advanced breast cancer.

In patients with some sub-type advanced breast cancer, neo-adjuvant chemotherapy combined with endocrine therapy may improve the pathological remission rate.

Premenopausal patients with triple negative breast caner and hormonal receptor positve breast cancer patients will be randominzed to have neoadjuvant chemotherapy combined with endocrine therapy or not.

DETAILED DESCRIPTION:
In this trial, patients with ER and or PR positive breast cancer will be separately randomized to have chemotherapy or chemotherapy combined with endocrine therapy according to their menstrual status. Letrozole for the postmenopausal women and ovarian function suppression for the premenopausal women. Patients with triple negative breast cancer will be randomized to have neoadjuvant chemotherapy combined with ovarian function suppression if she is premenopausal. Postermenopausal patients with triple negative breast caner will only have neoadjuvant chemotherapy.

Patients with Her2 overexpression can obtain anti-Her2 target therapy. This study has been amended to a 1:2 ratio to control and neoadjuvant chemotherapy combination of endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18years and ≤70 years;
2. At least on measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST). Histologically confirmed invasive breast cancer, tumor size ≥2 cm, T2-4 N0-3M0;
3. ER/PR/HER-2 and Ki-67 status detected on core biopsy. ER and/or PR positive was defined as >1% stained cells.HER2-positive is defined as immuno-histochemistry (IHC) 3+ or the ratio of HER2 gene signals to chromosome 17 signals >2.0 or HER2 gene copy >6.0.
4. No prior systemic or loco-regional treatment of breast cancer;
5. Adequate bone marrow function:WBC≥4.0×109/L, Absolute neutrophil count（ANC）≥1.5×109/L, Platelets（PLT）≥100×109/L, Hemoglobin（Hb）≥90g/L;aspartate aminotransferase(AST),Alanine aminotransferase (ALT)≤1.5 upper normal limit (UNL), creatinine≤1.5 UNL, bilirubin≤1.5UNL;
6. No obvious main organs dysfunction.

Exclusion Criteria:

1. Unwilling or unable to use an acceptable method of contraception in 8 weeks (including 8 weeks) after final dose of test drug;
2. Patient is pregnant or breast feeding;
3. Inflammatory breast cancer and metastatic breast cancer;
4. Any evidence of sense or motor nerve disorders;
5. Patients with medical conditions taht indicate intolerant to neoadjuvant therapy, including uncontrolled cardiovascular disease, severe infection;
6. Any concurrent malignancy other than breast cancer;
7. Know severe hypersensitivity to any drugs in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission rate | after 4 months preoperative treatment
  Pathological complete remission is defined as no invasive cancer in breast and axillary nodes.

SECONDARY OUTCOMES:
Number of Participants With Drug Related Treatment Adverse Events | 4 months during neoadjuvant therapy
  Adverse events that occurred on or after initial treatment that were absent before treatment or worsened during the treatment period relative to the pretreatment state.
Clinical and imaging response | 4 months during treatment
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests. (sonography, mammography, or MRI) after treatment
disease free survival (DFS) | 5 years
  DFS is defined as the time in months from randomization until first occurrence of locoregional recurrence, distant metastasis, contralateral breast cancer, second primary tumor, or death from any cause.
regional recurrence free survival (RRFS) | 5 years
  RRFS is defined as the time period between registration and first event
local recurrence free survival (LRFS) | 5 years
  LRFS is defined as the time period between registration and first event
overall survival (OS) | 5 years
  OS is defined as the time period between registration and first event
distant-disease- free survival (DDFS) | 5 years
  DDFS is defined as the time period between registration and first event
rate of tumor remission （RTR） | after 2 cycles and 4 cycles during neoadjuvant therapy
  RTR is defined as the proportion of tumor remission per unit time
serum markers | Pre-treatment and/or surgical
  Changes in the angiogenic serum markers(mirRNA, lncRNA, cirRNA), measured at diagnosis and surgery
molecular markers | Pre-treatment and/or surgical
  Pre-treatment and surgical expression of molecular markers （LHRHa receptor, EGFR，PD-L1)

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, Principal Investigator — RenJi Hospital
Locations (12):
- China (12):
  - Department of Thyroid and Breast Gland Surgery,Shenzhen Longgang Central Hospital, Shenzhen, Guangdong
  - HanDan Central Hospital, Handan, Hebei
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Department of Thyroid and Breast Surgery, The Affiliated Hospital of Inner Mongolia Medical Collage, Hohhot, Inner Mongolia
  - The second people's hospital of Kunshan city, Kunshan, Jiangsu
  - Department of Medical Oncology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality
  - Yueyang hospital of integrated traditional Chinese and Western medine, Shanghai, Shanghai Municipality
  - Armed Police Corps Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Department of Breast Surgery, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Zhoushan hospital, Zhoushan, Zhejiang

REFERENCES:
- [Derived] Wan C, Zhou L, Jin Y, Li F, Wang L, Yin W, Wang Y, Li H, Jiang L, Lu J. Strain ultrasonic elastography imaging features of locally advanced breast cancer: association with response to neoadjuvant chemotherapy and recurrence-free survival. BMC Med Imaging. 2023 Dec 21;23(1):216. doi: 10.1186/s12880-023-01168-2. PMID 38129778
- [Derived] Sun L, Yin W, Wu Z, Wang Y, Lu J. The Predictive Value of Pre-therapeutic Serum Gamma-glutamyl transferase in Efficacy and Adverse Reactions to Neoadjuvant Chemotherapy among Breast Cancer Patients. J Breast Cancer. 2020 Oct;23(5):509-520. doi: 10.4048/jbc.2020.23.e59. PMID 33154826
- [Derived] Bayarmaa B, Wu Z, Peng J, Wang Y, Xu S, Yan T, Yin W, Lu J, Zhou L. Association of LncRNA MEG3 polymorphisms with efficacy of neoadjuvant chemotherapy in breast cancer. BMC Cancer. 2019 Sep 5;19(1):877. doi: 10.1186/s12885-019-6077-3. PMID 31488093
- [Derived] Wu Z, Zhang L, Xu S, Lin Y, Yin W, Lu J, Sha R, Sheng X, Zhou L, Lu J. Predictive and prognostic value of ZEB1 protein expression in breast cancer patients with neoadjuvant chemotherapy. Cancer Cell Int. 2019 Mar 29;19:78. doi: 10.1186/s12935-019-0793-2. eCollection 2019. PMID 30976202